## The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Study 204981: A low interventional clinical study comparing error rates (critical and overall); between the ELLIPTA dry powder inhaler (DPI) and other DPIs, prior to any retraining in correct use, and as prescribed to treat COPD patients. |
|---|---|---|
| Compound Number | : | GSK573719+GW642444+GW685698 (GSK2834425) |
| Effective Date | : | 26-APR-2018 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be produced in the Clinical Study Report for Protocol 204981 (2016N301286\_00).
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

## RAP Author(s):

| Authors | | Date | Approval Method |
|---------------------|------------------------|------|-----------------|
| QSI. | tician ([Respiratory]) | N/A | N/A |
| Senior Program QSI. | mer ([Respiratory]) | N/A | N/A |

## The GlaxoSmithKline group of companies

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Statistics Leader, [Respiratory] (RD PCPS SPDS Clinical Statistics) | 26-APR-2018 | Pharma TMF |
| Clinical Development Scientist, [Respiratory] ([RD Respiratory HUP Clin Dev]) | 25-APR-2018 | Pharma TMF |
| Principal Clinical Data Manager, [Respiratory] ([RD PCPS Therapy Area Delivery) | 25-APR-2018 | Pharma TMF |
| Clinical Development Manager, [Respiratory] RD PCPS Therapy Area Delivery Resp 3 | 25-APR-2018 | Pharma TMF |
| SERM Manager, [Respiratory] RD<br>CMO GCSP SERM UK 3 | 25-APR-2018 | E-mail |
| Principal Statistician [Respiratory] (RD PCPS SPDS Clinical Statistics) | 25-APR-2018 | Pharma TMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| General Manager, Biostatistics and Programming ([Respiratory] QSI) | 25-APR-2018 | E-mail |
| Senior Manager, Biostatistics and Programming (Respiratory QSI) | 25-APR-2018 | E-mail |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | DDUCTION | 5 |
| 2. | CLIMIN | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Study Objective(s) and Endpoint(s) | |
| | 2.3. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| 3. | PLANI | NED ANALYSES | 15 |
| | 3.1. | Interim Analyses | 15 |
| | 3.2. | Final Analyses | 15 |
| 4. | ANAL` | YSIS POPULATIONS | |
| | 4.1. | Protocol Deviations | 16 |
| 5. | | IDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS | |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | | 5.4.1. Covariates and Other Strata | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling Conventions | 19 |
| 6. | | Y POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | |
| | | 6.1.1. Subject Disposition | |
| | | 6.1.2. Medical Conditions | |
| | | 6.1.3. Concomitant medication | 20 |
| 7. | | ACY ANALYSES | |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.5. Statistical Analyses / Methods | 21<br>21 |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | <mark>22</mark> |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.5. Statistical Analyses / Methods | |
| | | 7.2.5.1. Statistical Methodology Specification | |
| | 7.3. | Exploratory Efficacy Analyses | 24 |

| 8. | SAFETY | / ANALYSES | 26 |
|---|---|---|---|
| | 8.1. | Adverse Events Analyses | 26 |
| | 8.2. | Adverse Events of Special Interest | 26 |
| 9. | REFERI | ENCES | 27 |
| 10. | ADDENI | DICES | 20 |
| 10. | 10.1. | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population | |
| | 10.1. | Appendix 2: Schedule of Activities | |
| | 10.2. | 10.2.1. Protocol Defined Schedule of Events | |
| | 10.3. | Appendix 3: Study Phases and Treatment Emergent Adverse Events | |
| | 10.0. | 10.3.1. Study Phases | |
| | | 10.3.2. Treatment Phase Definitions | |
| | 10.4. | Appendix 4: Data Display Standards & Handling Conventions | |
| | | 10.4.1. Reporting Process | |
| | | 10.4.2. Reporting Standards | |
| | 10.5. | Appendix 5: Derived and Transformed Data | |
| | | 10.5.1. General | |
| | | 10.5.2. Study Population | 34 |
| | 10.6. | Appendix 6: Reporting Standards for Missing Data | |
| | | 10.6.1. Premature Withdrawals | 35 |
| | | 10.6.2. Handling of Missing Data | 35 |
| | | 10.6.2.1. Handling of Missing and Partial Dates | 35 |
| | 10.7. | Appendix 7: Abbreviations & Trade Marks | 37 |
| | | 10.7.1. Abbreviations | .37 |
| | | 10.7.2. Trademarks | |
| | 10.8. | Appendix 8: List of Data Displays | |
| | | 10.8.1. Data Display Numbering | |
| | | 10.8.2. Mock Example Shell Referencing | |
| | | 10.8.3. Deliverables | |
| | | 10.8.4. Study Population Tables | |
| | | 10.8.5. Efficacy Tables | |
| | | 10.8.6. Efficacy Figures | |
| | | 10.8.7. Safety Tables | |
| | | 10.8.8. ICH Listings | |
| | 40.0 | 10.8.9. Non-ICH Listings | |
| | 10.9. | Appendix 9: Example Mock Shells for Data Displays | .53 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronolog | jy: | |
|--------------------|-------------|----------|
| 2016N301286_00 | 24-JAN-2017 | Original |

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol.

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare the number of COPD patients making critical errors, when using their current prescribed inhaled medication, at V1 and prior to any re-training in correct use. | The percentage of participants making at least one critical error at V1 for each DPI tested. |
| Secondary Objectives | Secondary Endpoints The percentage of participants making at |
| To compare the number of COPD patients making overall errors, when using their current prescribed inhaled medication at V1 and prior to any re-training in correct use. | The percentage of participants making at least one overall error at V1 for each DPI tested. |
| To compare the number of COPD patients making critical and overall errors, when using their current prescribed inhaled medication at V2 (week 6). | <ul> <li>The percentage of participants making at least one critical error at V2 for each DPI tested.</li> <li>The percentage of participants making at least one overall error at V2 for each DPI tested.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| To explore, across all DPIs tested, if any association between critical errors, and key patient characteristics including: | Exploration of these characteristics will be investigated using a logistic regression model on the primary endpoint of the percentage of participants making at least one critical error at V1 for each inhaler tested, including each of these factors as terms in the model. • Age obtained from Demography. • Educational status from time in full time education. • Co-morbidities will be documented as relevant to DPI use. • Time on current DPI(s) and time since last trained will be documented categorically; however time on current DPI(s) will be included in the primary analysis model. |

| Objectives | Endpoints |
|---|---|
| Objectives | Level of control will be assessed by: COPD Assessment Test. Exacerbation History (Previous 1 year and required treatment with antibiotics and/or |
| | steroids). |

## 2.3. Study Design



## 2.4. Statistical Hypotheses

The primary purpose of this study is to assess the number of critical errors made by COPD patients for each DPI tested. The primary endpoint of the study is the percentage of participants making at least one critical error (critical error rate) for each DPI at V1. This will be analysed using logistic regression and will be adjusted for the covariate of time on current DPI.

For each DPI comparison:

- The null hypotheses are no difference between DPIs: H0: p1=p2
- The alternative hypothesis is that there is a difference between DPIs: HA: p1≠p2

## **Primary Endpoint**

The primary endpoint of the study is the percentage of participants making at least one critical error (critical error rate) for each DPI at V1

Table 1 Treatment groups

| Treatments | | Combination DPI Treatment Groups | | |
|---|---|---|---|---|
| Single DPI Treatment Groups | | ICS-LABA With<br>Spiriva HandiHaler<br>(LAMA) | | ICS-LABA With<br>Incruse ELLIPTA™<br>(LAMA) |
| Relvar ELLIPTA™ (ICS/LABA) A | | | G | |
| Symbicort Turbuhaler (ICS/LABA) B | | Н | | |
| Seretide DISKUS™ (ICS/LABA) C | | I | | |
| Spiriva HandiHaler (LAMA) D | | | | |
| Incruse ELLIPTA™ (LAMA) | | | | |
| Anoro ELLIPTA ™(LAMA/LABA) | | | | |
| Ultibro Breezhaler (LAMA/LABA) | | | | |
| Seebri Breezhaler (LAMA) | [ F | | | |

For this table the groups are referred to as treatment groups. For all other references in this RAP they will be referred to as *cohorts*.

## **Primary comparisons:**

- RELVAR ELLIPTA DPI vs. any other ICS/LABA (Seretide DISKUS™ or Symbicort Turbuhaler) DPI.
  - This comparison aims to compare critical error rates in the primary ICS/LABA DPIs.



- Group A versus group B
- Group A versus group C
- 2. INCRUSE ELLIPTA™ or ANORO ELLIPTA™ DPI vs. any other LAMA (Spiriva HandiHaler or Seebri Breezhaler), or LAMA/LABA (Ultibro Breezhaler) DPIs.
  - This comparison aims to compare critical error rates in the primary LAMA and LAMA/LABA DPIs.



- Group E versus Group D
- Group E versus Group F

## Other comparisons:

- 3. RELVAR ELLIPTA™ DPI vs. RELVAR ELLIPTA™ with any other LAMA (Spiriva HandiHaler or INCRUSE ELLIPTA™) DPI.
  - This aims to compare critical error rates in the primary DPI, simulating a triple therapy from one DPI (ELLIPTA) against triple therapy from two ELLIPTA DPIs, or from ELLIPTA DPI with any other LAMA DPI.



## Group A versus Group G

- RELVAR ELLIPTA™ DPI vs. all ICS/LABA (Seretide DISKUS™, RELVARELLIPTA™ or Symbicort Turbuhaler) DPIs with a LAMA (Spiriva HandiHaler, Seebri Breezhaler or INCRUSE ELLIPTA™) second DPI.
  - This aims to compare critical error rates in the primary DPI, simulating a triple therapy delivered in one ELLIPTA DPI against a triple therapy from any two other DPIs used in the study.



## Group A versus Group G+H+I

- 5. RELVAR ELLIPTA™ DPI with or without a LAMA DPI (Spiriva HandiHaler, Seebri Breezhaler or INCRUSE ELLIPTA™) vs. any other ICS/LABA (Seretide DISKUS™ or Symbicort Turbuhaler) DPI with or without a LAMA (Spiriva HandiHaler or Seebri Breezhaler) DPI.
  - This aims to compare critical error rates in the primary DPI, simulating a triple therapy delivered in one ELLIPTA DPI or combination of DPIs against a triple therapy using any other ICS/LABA delivering primary DPI.



- Group A+G versus B+H Group A+G versus C+I

Additionally, where there are 2 DPIs within a cohort, a further comparison will be made to compare the single DPI arm with the multiple DPI arm where errors from both devices are taken into consideration. See Table 2, Section 2.4.

These treatment comparisons above can be summarised in the following Table 2:

Table 2 Treatment comparisons

| Cohort: | Α | В | С | D | Е | F | G | Н | 1 |
|---|---|---|---|---|---|---|---|---|---|
| Primary device Secondary Device | Relvar<br>Ellipta | Symb<br>Turb | SFC<br>Diskus | Spiriva<br>HH | Inc. or<br>Anoro<br>Ellipta | Ultibro<br>or<br>Seebri<br>BH | (1) (1) Relvar Symb S | | |
| Primary Comparisons | | | | | | | | | |
| A vs B | Α | В | | | | | | | |
| A vs C | Α | | С | | | | | | |
| E vs D | | | | D | Е | | | | |
| E vs F | | | | | Е | F | | | |
| Other Comparisons | | | | | | | | | |
| A vs G (primary device) | А | | | | | | G1 | | |
| A v G<br>(both devices) | А | | | | | | G1/G2 | | |
| A vs G+H+I (primary device) | Α | | | | | | G1 | H1 | I1 |
| A vs G+H+I<br>(both devices) | А | | | | | | G1/G2 | H1/H2 | 11/12 |
| A+G vs B+H (primary device) | Α | В | | | | | G1 | H1 | |
| A+G vs B+H (both devices) | Α | В | | | | | G1/G2 | H1/H2 | |
| A+G vs C+I (primary device) | Α | | С | | | | G1 | | I1 |
| A+G vs C+I (both devices) | А | | С | | | | G1/G2 | | 11/12 |

Symb Turb: Symbicort Turbuhaler; SFC: Seretide; Inc.: Incruse; BH: Breezhaler;

HH: Handihaler

G1/G2 refers to errors in either primary device G1 or secondary device G2

H1/H2 refers to errors in either primary device H1 or secondary device H2

11/12 refers to errors in either primary device 11 or secondary device 12

#### **Secondary Endpoints**

The following secondary endpoints will be analysed in the same way as for the primary endpoint and using the same treatment comparisons:

- The percentage of participants making at least one overall error at V1 for each DPI tested.
- The percentage of participants making at least one critical error at V2 for each DPI tested.
- The percentage of participants making at least one overall error at V2 for each DPI tested.

For all formal statistical analyses where more than one DPI has been used, the comparison will be between the critical errors recorded on the primary DPI. Error rates will not be combined when dual DPIs are being used.

## **Exploratory Analysis**

The association between participants making at least one critical error (irrespective of the cohorts) and the key patient characteristics including age, educational Status, co-Morbidities (Arthritis (upper limbs), Neurological Disorders & Visual impairment), time on current DPI(s), time since last trained on DPI(s) and Level of control (CAT and Exacerbation History) will be examined at visit 1 for all the available subjects, irrespective of cohorts they belongs to.

# 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim Analysis planned

## 3.2. Final Analyses

All final planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Source database is locked and Data Management declare Source Data Lock.
- 5. Randomization codes have been distributed according to RandAllNG procedures.

  Note that this procedure will still be followed although the study is not formally randomized.
- 6. Database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

This study did not require formal randomisation to study treatment as subjects continued to use the maintenance medication they were already taking for COPD. However, in order to ensure that enrolment to treatment cohorts did not exceed the required number of subjects the study has implemented the use of RAMOS NG in order to monitor this. This also required that a randomisation was generated via RandallNG. The randomisation generated has a single treatment group (Own Treatment) and 9 strata levels (cohorts) for each of the treatment options detailed in Section 5.1 and Table 1 of the protocol.

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled (ASE) | Comprises of all participants who sign the ICF and for whom a record exists in the study database, including screen failures and any participant who was not screened but experienced an SAE between the date of informed consent and the planned date of the screening visit. | For subjects who do not enrol into a treatment group: Summary of study populations. Reason for screen failures Listing of SAEs |
| Randomised | All participants who were randomised. | No formal analysis will be performed on this population |
| Intent-To-Treat<br>(ITT) | All enrolled participants who have demonstrated use of their primary DPI. The population will be based on the treatment cohort to which the subject enrolled. Any subject who receives a treatment randomisation number will be considered to have been enrolled. | <ul><li>Study Population</li><li>Efficacy</li><li>Safety</li></ul> |
| Safety | This population will be the same as the ITT population. | |

#### NOTES:

 Please refer to Appendix 8: List of Data Displays which details the population to be used for each displays being generated.

## 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (PDMP).
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | | Combinations DPI Treatment Groups | |
|---|---|---|---|
| RandAll NG | | Data Displays for Reporting | |
| Code | Description | Description | Order in TFL |
| Α | Own Medication | Relvar Ellipta | 1 |
| В | Own Medication | Symbicort Turbuhaler | 2 |
| С | Own Medication | Seretide Diskus | 3 |
| D | Own Medication | Spiriva Handihaler | 4 |
| E | Own Medication | Incruse/Anoro Ellipta | 5 |
| F | Own Medication | Ultibro/Seebri Breezhaler | 6 |
| G | Own Medication | Relvar Ellipta + LAMA | 7 |
| Н | Own Medication | Symbicort Turbuhaler + LAMA | 8 |
| 1 | Own Medication | Seretide Diskus + LAMA 9 | |

#### NOTES:

- 1. Order represents treatments being presented in TFL, as appropriate.
- 2. Add a footnote to displays: LAMA = Spiriva Handihaler or Incruse Ellipta.

#### 5.2. Baseline Definitions

There are no baseline definitions to be defined.

## 5.3. Multicentre Studies

Data from all participating centres will be pooled prior to analysis.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

 The following is a list of covariates that will be used to explore, across all cohorts combined, if there is any association between critical errors and the key patient characteristic listed

| Category | Covariates and / or Subgroups |
|---|---|
| Age | 40-49; 50-59; 60-69; 70-79; 80+ years |
| Educational Status | 0-5; 6-10; 11-15; 16-20; 21+ years |
| Co-morbidities | Arthritis |
| | <ul> <li>Upper Limbs:(Shoulders, Elbows,</li> </ul> |
| | Hands/wrists/Fingers, Jaw and neck) |

| Category | Covariates and / or Subgroups |
|---|---|
| | Not upper limbs or No Arthritis (None, Back or lower body) Note:If both upper limbs and another location has been identified then the subject will be identified as upper limbs Visual impairment No visual impairment reported for either eye OR visual impairment in one eye only and marked as correctable OR visual impairment in both eyes and both eyes marked as correctable Vs Visual impairment in both eyes with neither or only |
| | 1 eye correctable OR Visual impairment in one eye which is not correctable. |
| | <ul> <li>Neurological Disorder</li> <li>Functional Disorder (Only current medical conditions) vs No Functional Disorder</li> </ul> |
| | <ul> <li>Dementia vs No Demintia</li> </ul> |
| | <ul> <li>Psychological Disorder vs. No psychological disorder</li> </ul> |
| Time since last trained on primary DPI | Categories are: • 3 months < x ≤ 6 months • 6 months < x ≤ 1 year |
| | <ul> <li>1 year &lt; x ≤ 2 years</li> <li>2 years &lt; x ≤ 3 years</li> <li>x &gt; 3 years</li> </ul> |
| Time on current primary DPI(s) | <ul> <li>Categories are: <ul> <li>3 months &lt; x ≤ 6 months</li> <li>6 months &lt; x ≤ 1 year</li> <li>1 year &lt; x ≤ 2 years</li> <li>2 years &lt; x ≤ 3 years</li> <li>x &gt; 3 years</li> </ul> </li> </ul> |
| Level of control | <ul> <li>CAT (&lt;10; &gt;=10)</li> <li>Exacerbation history in the prior year. (0, 1, ≥2 moderate/severe exacerbations in the prior year.</li> </ul> |

Note: If any visual impairment present and data doesn't exist whether it is correctable, then it is considered to be not-correctable

## 5.5. Multiple Comparisons and Multiplicity

There will be no adjustment for multiple comparisons on multiple endpoints in the analysis.

Given the exploratory nature of the study, multiplicity adjustments are not planned. There are 2 primary treatment comparisons. All other treatment comparisons are secondary.

## 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|--------------|--------------------------------------------------------------|
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| Section 10.2 | Appendix 2: Time & Events |
| Section 10.3 | Appendix 3: Treatment States and Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the ITT population, unless otherwise specified.

Study population displays including those of subject disposition, protocol deviations, demographic and baseline characteristics and prior and concomitant medications compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 8: List of Data Displays.

## 6.1.1. Subject Disposition

The study population summary will show the number of subjects overall who were enrolled, the number of screen failure and the number with each reason for screen failure, the number of subjects in each cohort and overall who were in the ITT population.

The end of study record summary shows the number of subjects who completed the study as well as the number who withdrew early from the study along with reasons for early withdrawal.

#### 6.1.2. Medical Conditions

The number and percentage of subjects reporting each current medical condition will be presented. This table will include a category of 'Cardiovascular Risk Factors'. All medical conditions must be summarised on this table regardless of frequency.

This will be repeated for past medical conditions.

#### 6.1.3. Concomitant medication

Non-COPD medications will be summarised by Anatomical-Therapeutic-Chemical (ATC) level 1 and ingredient. COPD medications will be summarised by Respiratory Medication Class (RMC) and will be derived for each COPD concomitant medication. Multi-ingredient medications will be presented according to their combination ATC classification rather than the classifications of the ingredients.

COPD and non-COPD medications will be listed separately.

A listing of the relationship between ATC Level 1, ingredient and verbatim text will be produced for non-COPD medications only.

## 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

The percentage of participants making at least one critical error at V1 for each DPI tested. See Table 2 (Section 2.4) for the cohort comparisons.

### 7.1.2. Summary Measure

Odds ratio at V1 for each of the comparisons detailed in Table 2 (Section 2.4).

## 7.1.3. Population of Interest

All subjects included in the ITT population.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

Subjects who have not performed the error assessment at V1 on their primary DPI will not form part of the ITT population (see Section 4).

There are no intercurrent events that impact treatment effect at V1. No missing data is anticipated at V1. There will be no imputation planned in the rare situation that subjects fail to complete an error assessment either in full or in part for one or both devices (where applicable).

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

The endpoint defined in Section 7.1.1 will be summarised using descriptive statistics, analysed as described in Section 7.1.5.1, graphically presented and listed.

## 7.1.5.1. Statistical Methodology Specification

## **Endpoint / Variables**

The proportion of non-responders (defined as making at least one critical error at V1). Non-response includes subjects where error assessment information is missing or incomplete at V1.

## **Model Specification**

- This endpoint will be analysed using logistic regression with treatment cohort as fixed effect
  and adjusting for the covariate of time on current primary DPI. All available data for all cohorts
  will be included in the model and pairwise treatment cohort comparisons for primary DPI vs
  primary DPI comparisons will be obtained from this model.
- In addition, a second model will be required in order to examine the pairwise treatment cohort comparisons for the dual device vs primary device comparisons.

## **Model Checking & Diagnostics**

Pearson residuals will be plotted for the model.

#### **Model Results Presentation**

• The odds ratio, 95% CI and p-value will be presented for the pairwise comparisons between DPIs/cohorts as detailed in Table 2 (Section 2.4). It will be based on a two-sided hypothesis testing approach of superiority.

## **Subgroup Analyses**

No subgroup analysis will be performed

#### **Sensitivity and Supportive Analyses**

No sensitivity analysis is planned for Primary endpoint

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

- The percentage of participants making at least one overall error at V1 for each DPI tested.
- The percentage of participants making at least one critical error at V2 for each DPI tested.
- The percentage of participants making at least one overall error at V2 for each DPI tested.

## 7.2.2. Summary Measure

For each of the endpoints detailed in 7.2.1 the summary measure is the odds ratio at the visit stated for each of the comparisons detailed in Table 2 (Section 2.4).

#### 7.2.3. Population of Interest

All subjects included in the ITT population.

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

Intercurrent events for secondary endpoint on visit 1 follow same handling method described in 7.1.4

The following intercurrent event is considered for V2;

Subject switches medication between V1 and V2

- New maintenance medication uses the same devices as previous maintenance medication at V1 and error assessments are performed on these new devices.
- New maintenance medication uses different devices to V1, but devices that are assessed in the study and for which error assessments are performed.
- New maintenance medication uses devices which are not being assessed in this study and thus no error assessment is available at V2.

For the purposes of this secondary endpoint analyses any error assessments following these events will be treated as missing. (i.e. if there are partial error assessments, the response will be

set to missing, or if there are full error assessments on alternative devices (or the same devices, but different medication) then these responses will also be set to missing)

Additionally, subjects may not provide an assessment at V2 for a number of reasons:

- Subject prematurely withdraws from the study before completing V2 assessments.
- For the treatment comparisons which take both devices into consideration (where applicable) a subject may have missed performing the assessment on the secondary device at V2.
- A subject may miss a component of a device assessment and all other question responses indicate correct use

For the purposes of these secondary analyses no imputation will be made for these missing scenarios.

In the situation where a subject may miss a component of a device assessment and one or more of the other question responses (critical error or overall error as applicable) indicate an error was made, then the subject would be a non-responder since the existing data already indicates this and the missing value has no additional impact on the response outcome.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 8: List of Data Displays and will be based on GSK data standards and statistical principles.

Endpoints defined in Section 7.2.1 will be summarised using descriptive statistics, analysed using appropriate statistical methods and graphically presented.

## 7.2.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

- The percentage of participants making at least one overall error at V1 for each DPI tested.
- The percentage of participants making at least one critical error at V2 for each DPI tested.
- The percentage of participants making at least one overall error at V2 for each DPI tested.

#### **Model Specification**

- These secondary endpoints will be analysed using logistic regression with treatment cohort as
  fixed effect and adjusting for the covariate of time on current primary DPI. All available data for
  all cohorts will be included in the model and pairwise treatment cohort comparisons for primary
  DPI vs primary DPI comparisons will be obtained from this model.
- A second model will be required in order to examine the pairwise treatment cohort comparisons for the dual device vs primary device comparisons.

#### **Model Checking & Diagnostics**

No model checking will be required for secondary endpoints.

#### **Model Results Presentation**

• The odds ratio, 95% CI and p-value will be presented for the pairwise comparisons between

DPIs/cohorts as detailed in Table 2 (Section 2.4). It will be based on a two-sided hypothesis testing approach of superiority.

### **Subgroup Analyses**

No subgroup analysis will be performed

#### **Sensitivity and Supportive Analyses**

- No sensitivity analysis is planned for these endpoints.
- If sufficient missing data warrants, a sensitivity analysis will be performed where the above scenarios are deemed to be non-responders.

# 7.3. Exploratory Efficacy Analyses

To explore, across all DPIs tested, if there is any association between critical errors, and key patient characteristics (Covariate or subgroups) including:

- Age.
- Educational Status.
- Co-Morbidities
  - Arthritis
  - Neurological Disorders
  - Visual impairment.
- Time on current DPI(s).
- Time since last trained on DPI(s).
- Level of control using the CAT.
- Exacerbation History.

The categories of interest for each of the covariates are described in Section 5.4.1.

For this analysis, all cohort data will be combined.

A summary table of errors will be produced for each patient characteristics.

Relationship of these characteristics will be investigated using a separate logistic regression model on the primary endpoint of the percentage of participants making at least one critical error and overall error at Visit 1 for each DPI tested, including each of these factors as terms in the model.

The interaction term between treatment cohort and characteristic will be added to the above model to investigate the interaction effect.

These analysis will be performed for each characteristic at a time. P-value from the first model and the interaction p-value from the second model will be produced for each characteristic adjusted seperately.

If any interaction is evident at the 10% significance level then further examination of the data may be performed in order to describe the interaction. It should be noted that due to the smaller groups of data and the number of tests, this investigation may highlight something which is a chance finding.

Graphical presentations of critical errors and overall errors for each patient characteristic will be produced.

## 8. SAFETY ANALYSES

The safety analyses will be based on the ITT population, unless otherwise specified.

## 8.1. Adverse Events Analyses

Adverse event summaries including the summary of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 8: List of Data Displays.

AE incidence will be summarised overall using the primary System Organ Class (SOC) and preferred term. All listings of AEs/SAEs will identify whether each adverse event occurred prestudy, during-study or post-study.

## 8.2. Adverse Events of Special Interest

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event.

Note: Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from on-going studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team agreements in place at the time of reporting.

A listing of subject numbers for individual adverse events of special interest will be produced along with a listing identifying all preferred terms which belong to each event of special interest.

The details of these planned displays are provided in Appendix 8: List of Data Displays.

## 9. REFERENCES

GlaxoSmithKline Document Number 2016N301286\_00, Protocol: An open-label, low interventional clinical study investigating error rates (critical and overall) prior to any retraining in correct use of the ELLIPTA dry powder inhaler (DPI) compared to other DPIs including; DISKUS, Turbuhaler, HandiHaler and Breezhaler as a monotherapy or in combination, in adult patients with Chronic Obstructive Pulmonary Disease (COPD), 24-January-2017.

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4: Analysis Populations | |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5: | General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Schedule of Activities |
| Section 10.3 | Appendix 3: Treatment States & Phases |
| Section 10.4 | Appendix 4: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.5 | Appendix 5: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Efficacy |
| Section 10.6 | Appendix 6: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Other RAP Appe | ndices |
| Section 10.7 | Appendix 7: Abbreviations & Trade Marks |
| Section 10.8 | Appendix 8: List of Data Displays |
| Section 10.9 | Appendix 9: Example Mock Shells for Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

A per protocol population is not defined for this study therefore there are no criteria leading to exclusion from a per protocol population. All deviations will be managed during the study according to the PDMP.

# 10.2. Appendix 2: Schedule of Activities

# 10.2.1. Protocol Defined Schedule of Events

| | Visit 0<br>Screening | Visit 1<br>Baseline | Visit 2 | Notes |
|---|---|---|---|---|
| | Day 1 (Can occur on same day as V1) | Day 1 (Can occur on same day as V0) | Week 6 ± 7 days | |
| Procedure | | | | |
| Screening (V0) | Х | | | Completed prior to V1 assessments. |
| Written informed consent | Х | | | V0 can take place on<br>the same day as V1. V1<br>should be completed no later<br>than 30 days after consent. |
| Participant demography | Х | | | Age, height, weight, year of birth, sex, ethnicity and geographic ancestry will be recorded. |
| Medical/disease history including COPD, smoking And Arthritis/Ophthalmic /Neurological history | X | | | Participant will have a medical history of COPD, smoking history, time on current DPI(s), time since last trained on DPI(s) and any comorbidities that may affect correct use of DPI recorded. |
| Exacerbation History | Х | | | Exacerbation history for previous year recorded. |
| COPD diagnosis | Х | | | Documented confirmation of COPD diagnosis from Physician. |
| Concomitant<br>medication<br>history including<br>COPD | Х | | | All current concomitant medication of relevance (Arthritic, Ophthalmic, Neurological medications) or related to an |

| | Visit 0<br>Screening | Visit 1<br>Baseline | Visit 2 | Notes |
|---|---|---|---|---|
| therapy history | | | | AE will be recorded. A minimum COPD therapy history for the preceding 2 years will be recorded. |
| Inclusion/exclusion criteria | Х | | | All criteria must be met prior to inclusion at V1. |
| Register the patient | Х | | | To ensure the correct number of patients are included on each arm. |
| CAT Score | Х | | | Take this for reference (exploratory). |
| Educational status | Х | | | No. of years spent in full time education. |
| Study Assessments<br>(V1<br>+V2) | | Х | Х | |
| Assess participant's ability to correctly use their DPI(s) and MDI(s) with Checklists | | Х | Х | No instruction provided by HCP before or during this assessment. |
| Correct use of DPI training | | Х | Х | Train participants should they make errors during demonstration |
| Adverse event/Serious adverse event assessment | | Х | Х | Collected until completion of study. |
| Prescriptions and health review | | Х | Х | Review changes in prescription and health between beginning and end of study. |

# 10.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

# 10.3.1. Study Phases

All data, where applicable, will be categorised according to the following treatment phases; prestudy, during- study and post- study. These definitions will be defined based on the date of Visit 1 and visit 2 given in the below table.

## 10.3.2. Treatment Phase Definitions

| Definition | Treatment Phase | | |
|---|---|---|---|
| Definition | Pre-study | During-study | Post-study |
| Before Visit 1 | Υ | | |
| Between V 1 and V 2 inclusive | | Υ | |
| After Visit 2 | | | Υ |

## 10.4. Appendix 4: Data Display Standards & Handling Conventions

## 10.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software and S-plus will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : gsk2834425\mid204981\final_01 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for the final_01 reporting effort. | |

## 10.4.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated: (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment (cohort) the subject belongs to.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.

#### Planned and Actual Time

- Reporting for tables, figures and formal statistical analysis:
  - Inhaler device errors nominal visit will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings if applicable (Refer to IDSL Statistical Principle 5.5.1).

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principles 7.01 to 7.13. | |

## 10.5. Appendix 5: Derived and Transformed Data

#### 10.5.1. General

## **Study Day**

- Calculated as the number of days from V1 Date
- Ref Date = Missing → Study Day = Missing
- Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
- Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

Note: Visit 1 date = Day 1

## **Study and Treatment Completion Definitions**

A participant is considered to have completed the study if he/she has completed all phases
of the study including the last scheduled procedure shown in the Schedule of Activities.

## 10.5.2. Study Population

#### Demography

#### Age

- Age will be calculated based on the Screening visit date (V0)
- Only year of birth is collected on the eCRF therefore day and month of birth are imputed as '30JUN' in order to derive age.
- Birth date will be presented in listings as 'YYYY'.

## **Body Mass Index**

• Calculated as weight (kg) / [height (m)]2

#### Subject disposition

#### **Treatment Compliance**

 Treatment compliance will not be calculated since no study treatment is dispensed in this study. Subjects are using their usual prescribed medication.

#### **COPD Exacerbation History**

- COPD exacerbation history is collected at visit 0/1. The eCRF collects the number of
  exacerbations in the unique categories of moderate or severe where a moderate COPD
  exacerbation is defined as an exacerbations that required treatment with systemic/oral
  corticosteroids and/or antibiotics (not involving hospitalization) and a severe COPD
  exacerbation is defined as an exacerbation that required in-patient hospitalization.
- Total number of moderate/severe COPD exacerbations for COPD exacerbation history are defined as the sum of moderate and severe COPD exacerbations for each subject.

# 10.6. Appendix 6: Reporting Standards for Missing Data

# 10.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completion of all phases of the study, including the last scheduled procedure shown in the schedule of activities.</li> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated by the use of a "blank" in subject listing. |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable", "Not evaluable" and "never trained on<br/>their DPI" are not considered to be missing data and should be displayed<br/>accordingly.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | <ul> <li>Start or end dates which are completely missing (i.e. no year specified) will remain missing, with no imputation applied.</li> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these result in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
## 10.7. Appendix 7: Abbreviations & Trade Marks

## 10.7.1. Abbreviations

| Abbreviation | Description |
|--------------|--------------------------------------------------------------|
| AE | Adverse Event |
| ASE | All Participants Enrolled |
| ATC | Anatomical Therapeutic Chemical Classification |
| CAT | COPD Assessment Test |
| COPD | Chronic Obstructive Pulmonary Disease |
| CRF | Case Report Form |
| DPI | Dry Powder Inhaler |
| GSK | GlaxoSmithKline |
| ICS | Inhaled Corticosteroid |
| IDSL | Integrated Data Standards Library |
| ITT | Intent-to-Treat |
| Kg | Kilogram |
| LABA | Long Acting β2-Agonist |
| LAMA | Long Acting Anticholinergic |
| m | Metre |
| MDI | Metered Dose Inhaler |
| MedDRA | Medical Dictionary for Regulatory Activities |
| PDMP | Protocol Deviation Management Plan |
| RAP | Reporting and Analysis Plan |
| RAMOS NG | Randomization & Medication Ordering System – Next Generation |
| RANDALLNG | GSK Randomization System – Next Generation |
| RMC | Respiratory Medication Class |
| RTF | Rich Text Format |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SoA | Schedule of Activities |
| SOC | System Organ Class |
| TFL | Tables, Figures & Listings |

## 10.7.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| ANORO ELLIPTA |
| INCRUSE ELLIPTA |
| RELVAR ELLIPTA |
| SERETIDE DISKUS |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| HandiHaler |
| SAS |
| Seebri Breezhaler |
| Spiriva Handihaler |
| Symbicort Turbuhaler |
| Ultibro Breezhaler |

### 10.8. Appendix 8: List of Data Displays

### 10.8.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|--------------|--------------|
| Study Population | 1.01 to 1.23 | N.A |
| Efficacy | 2.01 to 2.19 | 2.01 to 2.08 |
| Safety | 3.01 to 3.11 | N.A |
| Section | Listings | |
| ICH Listings | 1 to 16 | |
| Other Listings | 17 to 39 | |

### 10.8.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 9: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |

#### **NOTES:**

• Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.8.3. Deliverables

| Delivery | Description |
|----------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

## 10.8.4. Study Population Tables

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Populat | ion Analysed | | | | |
| 1.01 | ASE | IDSL_SP01 | Summary of Subject Populations | | SAC |
| 1.02 | ITT | POP_T1 | Summary of Attendance at Each Clinic Visit | Summarize for Screening, Visit1 and visit2 Summarize for Screening, Visit1 and visit2 Summarize for Screening, Visit1 and visit2Summarize for Screening, Visit 1 and Visit 2 | SAC |
| Subject | Disposition | | | | |
| 1.03 | ASE | IDSL_ES6 | Summary of Screening Status and Reasons for Screen Failures | Percentage for reason should be calculated based on number of screening failures refer Protocol Section 6.4 | SAC |
| 1.04 | ITT | IDSL_ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | SAC |
| 1.05 | ITT | IDSL_NS1 | Summary of Number of Subjects by Country and Centre | | SAC |
| 1.06 | ITT | IDSL_IE1 | Summary of Inclusion and Exclusion Criteria Deviations | | SAC |
| 1.07 | ITT | IDSL_DV1 | Summary of Important Protocol Deviations | | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demogr | aphic and Baseline ( | Characteristics | | | |
| 1.08 | ITT | IDSL_DM1 | Summary of Demographic Characteristics | Age category not required | SAC |
| 1.09 | ITT | IDSL_DM1 | Summary of Demographic Characteristics by Country | Age category not required: Page by country | SAC |
| 1.10 | ASE | IDSL_DM11 | Summary of Age Ranges | Categorise 18-64;65-84; >=85; Disclosure requirement | SAC |
| 1.11 | ITT | IDSL_DM5 | Summary of Race and Racial Combination | | SAC |
| 1.12 | ITT | IDSL_DM6 | Summary of Race and Racial Combinations details | | SAC |
| 1.13 | ITT | POP_T2 | Summary of COPD Duration at Screening | | SAC |
| 1.14 | ITT | POP_T3 | Summary of COPD Exacerbation History at Screening | | SAC |
| 1.15 | ITT | IDSL_FH1 | Summary of Family History of Cardiovascular Risk Factors | | SAC |
| 1.16 | ITT | IDSL_SU1 | Summary of Smoking History and Smoking Status at Screening | Include Years Smoked, Cigarettes/Day,<br>Smoking Pack Years*, Smoking Status<br>categories | SAC |
| 1.17 | ITT | POP_T4 | Summary of Baseline COPD Assessment Test (CAT) | For category refer Section 5.4.1 | SAC |
| 1.18 | ITT | IDSL_MH4 | Summary of Current Medical Conditions | | SAC |
| 1.19 | ITT | IDSL_MH4 | Summary of Past Medical Conditions | | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.20 | ITT | POP_T5 | Summary of Current Arthritis Location Details | | SAC |
| 1.21 | ITT | POP_T6 | Summary of Current Visual Impairment Details | | SAC |
| Prior an | Prior and Concomitant Medications | | | | |
| 1.22 | ITT | IDSL_CM1 | Summary of COPD Concomitant Medications | | SAC |
| 1.23 | ITT | IDSL_CM1 | Summary of Non-COPD Concomitant Medications | | SAC |

## 10.8.5. Efficacy Tables

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Primar | y Endpoint | | | | |
| 2.01 | ITT | EFF_T1 | Summary of Critical and Overall Errors | See shell for notes | SAC |
| 2.02 | ITT | EFF_T1 | Summary of Critical and Overall Errors by country | | SAC |
| 2.03 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one critical error at Visit 1 – Primary Device Comparisons | For comparisons of Primary devices Refer Section 2 Table 2 | SAC |
| 2.04 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one critical error at Visit 1 – Dual device vs Primary device Comparisons | For comparisons of Dual vs<br>Primary devices Refer Section 2<br>Table 2 | SAC |
| Secon | dary Endpoint | | | | |
| 2.05 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one overall error at Visit 1 – Primary Device Comparisons | For comparisons of Primary devices Refer Section 2 Table 2 | SAC |
| 2.06 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one overall error at Visit 1 – Dual device vs Primary device Comparisons | For comparisons of Dual vs<br>Primary devices Refer Section 2<br>Table 2 | SAC |
| 2.07 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one critical error at Visit 2 – Primary Device Comparisons | For comparisons of Primary devices Refer Section 2 Table 2 | SAC |
| 2.08 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one critical error at Visit 2 – Dual device vs Primary device Comparisons | For comparisons of Dual vs<br>Primary devices Refer Section 2<br>Table 2 | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.09 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one overall error at Visit 2 – Primary Device Comparisons | For comparisons of Primary devices Refer Section 2 Table 2 | SAC |
| 2.10 | ITT | EFF_T2 | Logistic Regression Analysis of percentage of Subjects making at least one overall error at Visit 2 – Dual device vs Primary device Comparisons | For comparisons of Dual vs<br>Primary devices Refer Section 2<br>Table 2 | SAC |
| Explor | atory Endpoint | | | | |
| 2.11 | ITT | EFF_T3 | Summary of Exploratory Subroups | Refer Section 5.4.1 | SAC |
| 2.12 | ITT | EFF_T4 | Summary of Subjects with at Least one Critical and Overall Error at Visit 1 by Age Group | Refer Section 5.4.1 for Age group | SAC |
| 2.13 | ITT | EFF_T4 | Summary of Subjects with at Least one Critical and Overall Error at Visit 1 by Educational Status Group | Refer Section 5.4.1 for Education status | SAC |
| 2.14 | ITT | EFF_T4 | Summary of Subjects with at Least one Critical and Overall Error at Visit 1 by Co-morbidities | Refer Section 5.4.1 for Comorbidities. | SAC |
| 2.15 | ITT | EFF_T4 | Summary of Subjects with at Least one of Critical and Overall Error at Visit 1 by Time Since Last Trained on Primary DPI | Refer Section 5.4.1 for time since last trained on primary DPI | SAC |
| 2.16 | ITT | EFF_T4 | Summary of Subjects with at Least one Critical and Overall Error at Visit 1 by Time on Current Primary DPI | Refer Section 5.4.1 for time on current primary DPI | SAC |
| 2.17 | ITT | EFF_T4 | Summary of Subjects with at Least one Critical or Overall Error at Visit 1 by Level of Control | Refer Section 5.4.1 for time on current primary DPI for level of control – this includes both CAT and Exac history | SAC |

| Efficac | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18 | ITT | EFF_T6 | Exploratory Analysis of Patient Characteristics and Interaction with Cohort using Logistic Regression for Critical Error and Overall Errors at Visit 1 | | SAC |
| Additional Tables | | | | | |
| 2.19 | ITT | EFF_T1 | Summary of Rescue MDI Critical and Overall Errors | | SAC |

## 10.8.6. Efficacy Figures

| Efficac | y: Figures | | | | | |
|---|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] | |
| 2.01 | ITT | EFF_F1 | Percentage of Subjects with at Least One critical Error | Present both visit 1 and visit 2 on the same panel | SAC | |
| 2.02 | ITT | EFF_F1 | Percentage of Subjects with at Least One Overall Error | ercentage of Subjects with at Least One Overall Error Present both visit 1 and visit 2 on the same panel | | |
| 2.03 | ITT | EFF_F2 | Percentage of Subjects with at Least One Critical Error and Overall Error at Visit 1 – by Age group | | | |
| 2.04 | ITT | EFF_F2 | Percentage of Subjects with at Least One Critical Error and Overall Error at Visit 1 – by Educational Status Group Present critical and overall in side by side plots on the same page | | Percentage of Subjects with at Least One Childar Effor and I side by side plots on | SAC |
| 2.05 | ITT | EFF_F2 | Percentage of Subjects with at Least One Critical Error and Overall Error at Visit 1 – by Comorbidity group | Present critical and overall in side by side plots on the same page, page by each comorbidity (Arthritis, Visual Impairment, Neurological) | SAC | |
| 2.06 | ITT | EFF_F2 | Percentage of Subjects with at Least Critical Error and Overall Error at Visit 1 – by Time Since Last Trained on Primary DPI | Present critical and overall in side by side plots on the same page | SAC | |
| 2.07 | ITT | EFF_F2 | Percentage of Subjects with at Least One Critical Error and Overall Error at Visit 1 – by Time on Current Primary DPI | Present critical and overall in side by side plots on the same page | SAC | |

| Efficac | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.08 | ITT | EFF_F2 | Percentage of Subjects with at Least One Critical Error and Overall Error at Visit 1 – by Level of Control | Present critical and overall in side by side plots on the same page. | SAC |

## 10.8.7. Safety Tables

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | o. Population IDSL / Example Shell | | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.01 | ITT | IDSL_AE13 | Overview of Adverse Events | | SAC |
| 3.02 | ITT | IDSL_AE1 | Summary of During-Study Adverse Events by System<br>Organ Class and Preferred Term | | SAC |
| 3.03 | ITT | IDSL_AE1 | Summary of Post-Study Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.04 | ITT | IDSL_AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | Include Serious, Drug-Related<br>Serious, Fatal and Drug-Related<br>Serious | SAC |
| 3.05 | ITT | IDSL_AE1 | Summary of During-Study Serious Adverse Events by System Organ Class and Preferred Term | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.06 | ITT | IDSL_AE1 | Summary of During-Study Fatal Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.07 | ITT | IDSL_AE1 | Summary of During-Study Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.08 | ITT | IDSL_AE1 | Summary of During-Study Drug-related Fatal Serious<br>Adverse Events by System Organ Class and Preferred<br>Term | | SAC |
| 3.09 | ITT | IDSL_AE15 | Summary of During-study Common (>=3% in Either Cohort) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | SAC |
| Serious | s and Other Sig | nificant Adver | se Events | | |
| 3.10 | ITT | IDSL_AE1 | Summary of During-Study Non-Fatal Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 3.11 | ITT | IDSL_AE1 | Summary of During-Study Adverse Events Leading to Permanent Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | | SAC |

## 10.8.8. ICH Listings

| ICH: L | istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | 1 | | | |
| 01 | ASE | IDSL_ES7 | Listing of Reasons for Screen Failure | | SAC |
| 02 | ITT | IDSL_ES2 | Listing of Reasons for Study Withdrawal | Followup columns are not needed | SAC |
| Protoc | ol Deviations | | | | |
| 03 | ITT | IDSL_DV2 | Listing of Important Protocol Deviations | | SAC |
| 04 | ITT | IDSL_IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Demo | graphic and Basel | ine Characterist | ics | | |
| 05 | ITT | IDSL_DM2 | Listing of Demographic Characteristics | Include BMI in the listing | SAC |
| 06 | ITT | IDSL_DM9 | Listing of Race | | SAC |
| Advers | se Events | | | | |
| 07 | ASE | IDSL_AE8 | Listing of All Adverse Events | | SAC |
| 08 | ITT | IDSL_AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 09 | ITT | IDSL_AE8 | Listing of Non-Fatal Adverse Events | | SAC |
| 10 | ITT | IDSL_AE8 | Listing of Fatal Adverse Events | | SAC |

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 11 | ITT | IDSL_AE2 | Listing of Relationship Between Adverse Event<br>System Organ Class, Preferred Term and Verbatim<br>Text | | SAC |
| Seriou | s and Other Signif | icant Adverse E | vents | | |
| 12 | ITT | IDSL_AE8 | Listing of Fatal Serious Adverse Events | | SAC |
| 13 | ITT | IDSL_AE8 | Listing of Non-Fatal Serious Adverse Events | | SAC |
| 14 | ITT | IDSL_AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| Inhaler | errors | | | | |
| 15 | ITT | EFF_L1 | Listing of Inhaler Used at Visit 1 and Visit 2 | | SAC |
| 16 | ITT | EFF_L2 | Listing of Subject Errors | | SAC |

## 10.8.9. Non-ICH Listings

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subje | ct Population | | | | |
| 17 | ITT | POP_L1 | Listing of Subjects by Country and Centre | | SAC |
| 18 | ITT | POP_L2 | Listing of Family History of Cardiovascular Risk Factors at Screening | | SAC |
| 19 | ITT | POP_L3 | Listing of COPD Duration at Screening | | SAC |
| 20 | ITT | POP_L4 | Listing of Smoking History and Smoking Status at Screening | | SAC |
| 21 | ITT | POP_L5 | Listing of COPD Assessment Test (CAT) at Screening | | SAC |
| 22 | ITT | POP_L6 | Listing of Current Arthritis Location details | | SAC |
| 23 | ITT | POP_L7 | Listing of Visual Impairment details | | SAC |
| Medica | al Conditions | | | | • |
| 24 | ITT | IDSL_MH2 | Listing of Medical Conditions | | SAC |

| Non-IC | CH: Listings | | | |
|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Programming Notes | Deliverable<br>[Priority] |
| Conco | mitant Medicati | ons | | |
| 25 | ITT | IDSL_CM3 | Listing of COPD Concomitant Medications | SAC |
| 26 | ITT | IDSL_CM3 | Listing of Non-COPD Concomitant Medications | SAC |
| 27 | ITT | IDSL_CM6 | Relationship between ATC Level 1, Ingredient and Verbatim Text for non-COPD medications | SAC |
| Advers | e Events of Sp | ecial Interest | | |
| 28 | ITT | SAFE_L1 | Listing of Subject Numbers for Individual Adverse<br>Events of Special Interest | SAC |
| 29 | ITT | SAFE_L2 | Listing of Adverse Event of Special Interest Group,<br>Subgroup, Sub-SMQ and Preferred Term | SAC |

| Non-le | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / Example<br>Shell | Title | Deliverable<br>[Priority] | |
| Cardio | ovascular Event | s (Patient profiles) | | | • |
| 30 | ASE | IDSL_ CVEND1 | Lisiting of Arrhythmias | | SAC |
| 31 | ASE | IDSL_ CVEND2 | Lisiting of Congestive Heart Failure | | SAC |
| 32 | ASE | IDSL_ CVEND3 | Lisiting of Cerebrovascular Events Stroke (CVA) and Transient Ischemic Attack (TIA) | | SAC |
| 33 | ASE | IDSL_ CVEND4 | Lisiting of Deep Vein Thrombosis (DVT)/Pulmonary Embolism (PE) | | SAC |
| 34 | ASE | IDSL_ CVEND5 | Lisiting of Myocardial Infarction/Unstable Angina | | SAC |
| 35 | ASE | IDSL_ CVEND6 | Lisiting of Peripheral Arterial Thromboembolism | | SAC |
| 36 | ASE | IDSL_ CVEND7 | Lisitng of Pulmonary Hypertension | | SAC |
| 37 | ASE | IDSL_ CVEND8 | Lisiting of Revascularisation | | SAC |
| 38 | ASE | IDSL_ CVEND9 | Listing of Valvulopathy | | SAC |
| 39 | ASE | IDSL_DEATH | Listing of All cause deaths | | SAC |

## 10.9. Appendix 9: Example Mock Shells for Data Displays

POP\_T1


Population: Intent-to-Treat

Table 1.x
Summary of Attendance at Each Clinic Visit

| Visit | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | Cohort D<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|---|
| Screening | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Visit1 | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Visit2 | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |

Note: Display Cohort name given in the section 5

POP\_T2

Protocol: 204981

Population: Intent-to-Treat


Table 1.x
Summary of COPD Duration at Screening

| | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Duration of COPD | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| < 6 months | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 6 months to < 1 year | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 5 years to < 10 years | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 10 years to < 15 years | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 15 years to < 20 years | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 20 years to < 25 years | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >= 25 years | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| COPD Type | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Chronic bronchitis | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Emphysema | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Display Cohort name given in the section 5

POP\_T3

Protocol: 204981

Population: Intent-to-Treat


Table 1.x Summary of COPD Exacerbation History at Screening

| | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Moderate COPD exacerbations | | | | | | |
| n<br>0<br>1<br>>=2 | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) | xxx<br>xxx (xx%)<br>xxx (xx%)<br>xxx (xx%) |
| Severe COPD exacerbations | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=2 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Total number of moderate/severe COPD exacerbations | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| 0 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| 1 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=2 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Display Cohort name given in the section 5

POP\_T4

Protocol: 204981

Population: Intent-to-Treat


Table 1.x
Summary of Baseline COPD Assessment Test (CAT)

| | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| CAT Score | | | | | | |
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Min. | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |
| Q1 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q3 | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Max. | Xxx | Xxx | Xxx | Xxx | Xxx | Xxx |
| CAT Category | | | | | | |
| n | XXX | Xxx | XXX | XXX | XXX | XXX |
| < 10 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| >=10 | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Note: Display Cohort name given in the section 5

POP\_T5


Population: Intent-to-Treat

Table 1.x Summary of Current Arthritis Location Details

| | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| Current Arthritis | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Arthritis Location | | | | | | |
| Back | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Neck | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Shoulders | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Elbows | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Hands, Wrists and fingers | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Lower body | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Jaw | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

#### Footnote:

Subjects may have more than one Arthritis location, so percentages may sum to more than 100%.

Percentage for Current Arthritis are calculated based on number of subjects in each Cohort.

Percentage for Arthritis Location are calculated based on number of subjects having Current Athritis

Note: Display Cohort name given in the section 5

POP\_T6


Population: Intent-to-Treat

Table 1.x Summary of Current Visual Impairment Details

| | Cohort A<br>(N=XXX) | Cohort B<br>(N=XXX) | Cohort C<br>(N=XXX) | | Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|---|---|
| n | XXX | XXX | XXX | XXX | XXX | XXX |
| Left eye | | | | | | |
| Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Not- Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Right eye | , , | , , | , , | | , , | , , |
| Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Not- Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Both eyes | , , | , , | , , | | , , | , , |
| Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Not- Correctable | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |
| Correctable in only one eye | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) | xxx (xx%) |

Footnote:

[1] Percentage is calculated based on number of subjects having visual Impairment (n)

Note: Display Cohort name given in the section 5


#### CONFIDENTIAL

EFF\_T1

Protocol: 204981

Population: Intent-to-Treat

#### Table 2.01 Summary of Critical and Overall Errors

Cohort : A (N=XXX)
Device: Ellipta

| Inhaler errors test | Visit 1 | Visit 2 |
|---|---|---|
| N | XX | XX |
| Number of Subjects with at least one Error<br>Number of Subjects with at least one Critical Error | XX (XX%)<br>XX (XX%) | XX (XX%)<br>XX (XX%) |
| Total Number of Errors Total Number of Critical Errors | XX<br>XX | XX<br>XX |
| Failed to open cover [1] Inhalation manoeuvre: long, steady, deep Blocked air inlet during inhalation manoeuvre Shook the device after dose preparation [1] No exhalation before an inhalation Exhaled directly into mouthpiece [1] No seal by the lips round the mouthpiece during the inhalation [1] Did not hold breath Did not close the device (Note: this is an error but one which | XX (XX%) | XX (XX%) |

<sup>[1]</sup> Indicates a Critical Error.

Note: Percentages for number of subjects with at least one error are calculated from the total number of subjects who used the device(s)

Note: Percentages for type of errors are calculated from the number of subjects with overall errors.

Repeat for each cohort. Within those cohorts with 2 devices, produce 3 pages, 1st page with the first 4 lines above, 2nd page with the primary device errors (in the same way as above) and 3rd page with the second device errors (as above). (i.e. see the error table in '215 for the treatment arms with multiple devices)

Also note that the device page heading should be the device alone and not the drug, the drug will be evident from the cohort label.

EFF\_T2


Population: Intent-to-Treat

Table 2.xx
Logistic Regression Analysis of percentage of Subjects making at least one critical error at Visit 1 – Primary Device Comparisons

| Cohort | N | n | Critical Error | Zero Critical Error | 0.R. | 95% C.I. | p-value |
|---|---|---|---|---|---|---|---|
| Α | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| В | XX | XX | xx (xx%) | xx (xx%) | | | |
| Α | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| С | XX | XX | xx (xx%) | xx (xx%) | | | |
| Е | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| D | XX | XX | xx (xx%) | xx (xx%) | | , | |
| Е | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| F | XX | XX | xx (xx%) | xx (xx%) | | , | |
| Α | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| G1 | XX | XX | xx (xx%) | xx (xx%) | | | |
| Α | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| G1+H1+I1 | XX | XX | xx (xx%) | xx (xx%) | | , | ` |
| A+G1 | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| B+H1 | XX | XX | xx (xx%) | xx (xx%) | | , | |
| A+G1 | XX | XX | xx (xx%) | xx (xx%) | X.XXX | (x.xxx,x.xxx) | X.XXX |
| C+I1 | XX | XX | xx (xx%) | xx (xx%) | | , , | |

Note: Display Cohort name instead of Cohort codes

EFF\_T3 Protocol: 204981 Page 1 of x

Population: Intent-to-Treat

Table 1.x Summary of Exploratory Subgroups

| Covariates and / or Subgroups | Cohort A<br>(N=XX) | Cohort B<br>(N=XX) | <br>Cohort I<br>(N=XXX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| Age | , | , , | | |
| 40-49 Years | XXX | XXX | XXX | XXX |
| 50-59 years | XXX | XXX | XXX | XXX |
| 60-69 years | XXX | XXX | XXX | XXX |
| 70-79 years | XXX | XXX | XXX | XXX |
| >=80 years | XXX | XXX | XXX | XXX |
| Educational status | | | | |
| 0-5 years | XXX | XXX | XXX | XXX |
| 6-10 years | XXX | XXX | XXX | XXX |
| 11-15 years | XXX | XXX | XXX | XXX |
| 16-20 years | XXX | XXX | XXX | XXX |
| >=21 years | XXX | XXX | XXX | XXX |
| Arthritis | | | | |
| Upper Limbs | XXX | XXX | XXX | XXX |
| Not upper limbs or No Arthritis | XXX | XXX | XXX | XXX |
| Visual Impairment | | | | |
| Visual Impairment not correctable | XXX | XXX | XXX | XXX |
| Visual Impairment correctable / No Visual | XXX | XXX | XXX | XXX |
| Impairment | | | | |
| Neurological disorder | | | | |
| Functional disorder | XXX | XXX | XXX | XXX |
| No functional disorder | XXX | XXX | XXX | XXX |
| Dementia | XXX | XXX | XXX | XXX |
| No dementia | XXX | XXX | XXX | XXX |
| Psychological disorder | XXX | XXX | XXX | XXX |

## 2018N371346\_00 204981

| No psychological disorder | XXX | XXX | XXX | XXX |
|----------------------------------------|-----|-----|-----|-----|
| Time since last trained on primary DPI | | | | |
| >3 to ≤ 6 Months | XXX | XXX | XXX | XXX |
| >6 Months to ≤ 1 Year | XXX | XXX | XXX | XXX |
| >1 year to ≤ 2 Years | XXX | XXX | XXX | XXX |
| >2 Years to ≤ 3 Years | XXX | XXX | XXX | XXX |
| > 3 Years | XXX | XXX | XXX | XXX |
| Time on current primary DPI(s) | | | | |
| >3 to ≤ 6 Months | XXX | XXX | XXX | XXX |
| >6 Months to ≤ 1 Year | XXX | XXX | XXX | XXX |
| >1 year to ≤ 2 Years | XXX | XXX | XXX | XXX |
| >2 Years to ≤ 3 Years | XXX | XXX | XXX | XXX |
| > 3 Years | XXX | XXX | XXX | XXX |
| COPD Assessment test (CAT) | | | | |
| <10 | XXX | XXX | XXX | XXX |
| >=10 | XXX | XXX | XXX | XXX |
| Exacerbation history in Prior year | | | | |
| 0 | XXX | XXX | XXX | XXX |
| 1 | XXX | XXX | XXX | XXX |
| >=2 | XXX | XXX | XXX | XXX |

EFF\_T4

Protocol: 204981

Population: Intent-to-Treat


Table 2.XX Summary of Critical and Overall Errors at Visit 1 by Age Group

| Age Group | Ν | n | Critical Error | Overall Error |
|-------------|----|----|----------------|---------------|
| 40-49 Years | XX | XX | XX (XX%) | XX (XX%) |
| 50-59 years | XX | XX | XX (XX%) | XX (XX%) |
| 60-69 years | Xx | XX | XX (XX%) | XX (XX%) |
| 70-79 years | Xx | XX | XX (XX%) | XX (XX%) |
| >=80 years | Xx | XX | XX (XX%) | XX (XX%) |

EFF\_T5


Population: Intent-to-Treat

Table 2.xx
Exploratory Analysis of Patient Characteristics and Interaction with Cohort using Logistic Regression for Critical Error and Overall Errors at Visit 1

| | | | | Interaction | with Cohort |
|---|---|---|---|---|---|
| | | Critical Error | Overall Error | Critical Error | Overall Error |
| Covariates and / or Subgroups | Category | p-value | p-value | p-value | p-value |
| Age: | 40-49 years<br>50-59 years<br>60-69 years<br>70-79 years<br>>=80 years | X.XXX | X.XXX | X.XXX | X.XXX |
| Educational status | 0-5 years<br>6-10 years<br>11-15 years<br>16-20 years<br>>=21 years | X.XXX | X.XXX | X.XXX | X.XXX |
| Arthritis | Yes/ No | X.XXX | X.XXX | X.XXX | X.XXX |
| Visual Impairment | Yes/ No | X.XXX | X.XXX | X.XXX | X.XXX |
| Functional disorder | Yes/ No | X.XXX | X.XXX | X.XXX | X.XXX |
| Dementia | Yes/ No | X.XXX | X.XXX | X.XXX | X.XXX |
| Psychological disorder | Yes/ No | X.XXX | X.XXX | X.XXX | X.XXX |
| Time since last trained on primary DPI | >3 to ≤ 6 Months<br>>6 Months to ≤ 1 Year<br>>1 to ≤ 2 Yearrs;<br>>2 to ≤ 3 Years;<br>> 3 Years | X.XXX | X.XXX | X.XXX | X.XXX |
| Time on current primary DPI(s) | _ " _ | X.XXX | X.XXX | X.XXX | X.XXX |

| $\sim$ | | | ΝТ | A I |
|--------|-----|-----|-------|-----|
| CO | IVE | IDE | N 1 1 | AL |

2018N371346\_00 

| COPD Assessment test (CAT). | <10/>=10 | X.XXX | X.XXX | X.XXX | X.XXX |
|-----------------------------|----------|-------|-------|-------|-------|
| Exacerbation history | 0,1, ≥2 | X.XXX | X.XXX | X.XXX | X.XXX |

EFF\_F1

Protocol: 204981

Population: Intent to Treat


Figure X.X
Percentage of Subjects with at Least One Critical Error



Programming note: Please present Cohort names instead of Cohort Codes. Please use different pattern for diifernt visit.

Footnote: For the cohort with two devices (G,H and I), the critical error is counted only for primary devices.

EFF\_F2


Population : Intent to Treat

Figure X.X
Percentage of Subjects with at Least One Critical and Overall Error
By Age Group



AGE GROUP

.Repeat for other exploratory covariates groups of interest

POP\_L1

Protocol: 204981

Population: Intent-to-Treat


# Listing xx Listing of Subjects by Country and Centers

| Country | Inv. at Centre | Investigator<br>Name<br> | Subject | Cohort |
|---|---|---|---|---|
| Netherlands | PPD | | | DISKUS + HandiHaler |
| | | | | ELLIPTA/DISKUS + HandiHaler |
| | | | | DISKUS + HandiHaler/ELLIPTA |
| United Kingdom | | | | DISKUS + HandiHaler |
| | | | | ELLIPTA/DISKUS + HandiHaler |

POP\_L2


Population: Intent-to-Treat

## Listing xx Listing of Family History of Cardiovascular Risk Factors at Screening

| Inv. at Centre | Subject | Cohort | Family History [1] |
|---|---|---|---|
| PPD | | DISKUS + HandiHaler/ELLIPTA/Q1 | Yes |
| | | ELLIPTA/DISKUS + HandiHaler/Q1 | Unknown |
| | | DISKUS + HandiHaler/ELLIPTA/Q2 | Unknown |
| | | ELLIPTA/DISKUS + HandiHaler/Q2 | Yes |
| | | DISKUS + HandiHaler/ELLIPTA/Q2 | Unknown |

Footnote: [1] Family history of premature coronary artery disease in women < 65 years or men < 55 years in first degree relatives only (e.g., biological mother or father, biological brother or sister, biological son or daughter).

POP\_L3


Population: Intent-to-Treat

Listing xx
Listing of COPD Duration at Screening

| Inv. at Ce | ntre Sul | bject | Cohort | Duration |
|---|---|---|---|---|
| PPD | | | DISKUS + HandiHaler/ELLIPTA/Q1 | >=1 year to <5 years |
| | | | ELLIPTA/DISKUS + HandiHaler/Q1 | >=10 years to <15 |
| | | | Years | |
| | | | DISKUS + HandiHaler/ELLIPTA/Q2 | >=1 year to <5 years |
| | | | ELLIPTA/DISKUS + HandiHaler/Q2 | >=5 years to <10 |
| | | | Years | |
| | | | DISKUS + HandiHaler/ELLIPTA/Q2 | >=1 year to <5 years |

POP\_L4

Population: Intent-to-Treat

Listing xx
Listing of Smoking History and Smoking Status at Screening

| Inv. at centre | Subject | Cohort | Years Smoked | Cigarettes<br>per day | Smoking Pack Years [1] | Smoking status |
|---|---|---|---|---|---|---|
| PPD | | DISKUS +<br>HandiHaler/ELLIPTA/Q1 | 25 | 20 | 25 | Former Smoker |
| | | ELLIPTA/DISKUS +<br>HandiHaler/Q1 | 50 | 30 | 75 | Current Smoker |
| | | DISKUS +<br>HandiHaler/ELLIPTA/Q2 | 50 | 15 | 38 | Former Smoker |
| | | ELLIPTA/DISKUS +<br>HandiHaler/Q2 | 26 | 20 | 26 | Never Smoked |

POP\_L5


Population: Intent-to-Treat

## Listing xx Listing of COPD Assessment Test (CAT) at Screening

| Inv. at Centre | Subject | Cohort<br>DISKUS + HandiHaler/ELLIPTA/Q1 | CAT Total Score<br>15 |
|---|---|---|---|
| | | ELLIPTA/DISKUS + HandiHaler/Q1 | 10 |
| | | DISKUS + HandiHaler/ELLIPTA/Q2 | 10 |
| | | ELLIPTA/DISKUS + HandiHaler/Q2 | 16 |

2018N371346\_00 204981

POP\_L6

Protocol: 204981

Population: Intent-to-Treat


## Listing xx Listing of Current Arthritis Location Details



204981

CONFIDENTIAL

POP\_L7

Page 1 of x Protocol: 204981 Population: Intent-to-Treat

Listing xx Listing of Visual Impairment Details

| Inv. at Centre | Subject | Cohort | Eyes affected | Eyes corrected |
|---|---|---|---|---|
| PPD | | DISKUS + HandiHaler/ELLIPTA/Q1 | Left | Left |
| | | ELLIPTA/DISKUS + HandiHaler/Q1 | Right | Right |
| | | DISKUS + HandiHaler/ELLIPTA/Q2 | Left | Left |
| | | ELLIPTA/DISKUS + HandiHaler/Q2 | Both | Right |
| | | DISKUS + HandiHaler/ELLIPTA/Q2 | Both | Both |

2018N371346\_00 204981

### EFF\_L1

Protocol: 204981

Population: Intent-to-Treat


## Listing xx

Listing of Inhaler Use at Visit 1 and Visit 2

| Inv. at centre | Subject |
|----------------|---------|
| PPD | |

Visit 1 Relvar Ellipta + Spirivia HandiHaler Relvar Ellipta

Relvar Ellipta

Visit 2 Relvar Ellipta

Relvar Ellipta

Switched the device/ medication Y

Relvar Ellipta+Other

Υ

Inhalation

EFF\_L2

Protocol: 204981

Population: Intent-to-Treat


Listing xx Listing of Critical and Overall Inhaler Errors

| Inv. at centre | Subject | Cohort<br>DISKUS +<br>HandiHaler | Actual<br>Cohort<br>DISKUS +<br>HandiHaler | Visit<br>Visit 1 | Total<br>3 | Device<br>HandiHaler | Type of Error<br>Capsule did not rattle [1] |
|---|---|---|---|---|---|---|---|
| | | | | | | | Inhalation manoeuvre: was slow, deep |
| | | | | | | DISKUS | No exhalation before an |

Footnote: [1] Indicates a Critical Error.

Programming note: The number in total column displays number of errors the subject had made irrespective of devices. Cohort and Actual Cohort are trtgrp and atrtgrp.

List only the error assessment not completed correctly under "Type of error" column.

SAFE\_L1


Population: Intent-to-Treat

Listing xx
Listing of Subject Numbers for Individual Adverse Events of Special Interest

AESI Group: CV effects/Hypertension (SMQ)

| System Organ Class Preferred Term | Treatment | No.<br>with<br>Event | Subject |
|---|---|---|---|
| Investigations Blood pressure increased | DISKUS + HandiHaler | 1 | PPD |
| Vascular disorders<br>Hypertension | DISKUS + HandiHaler | 2<br>1 | |

SAFE\_L2

Protocol: 204981


Population: Intent-to-Treat

Listing xx
Listing of Adverse Event of Special Interest Group, Subgroup, Sub-SMQ and Preferred Term

AESI Group

AESI Subgroup

Sub-SMQ

Preferred Term

Adrenal suppression

-----

ACTH stimulation test abnormal Addison's disease

Adrenal androgen deficiency

Adrenal atrophy
Adrenal insufficiency